CLINICAL TRIAL: NCT01626521
Title: Value of Prothrombin Fragment F1+2 in the Diagnosis of Pulmonary Embolism in Patients With Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0033-12-HYMC
Record Dates: First submitted 2012-06-17; First posted 2012-06-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Embolism | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD Exacerbation: Patients admitted to hospital with COPD exacerbation
  Interventions: Other: CT pulmonary angio, blood tests

INTERVENTIONS:
Other: CT pulmonary angio, blood tests — CT pulmonary angiography to determine PE and laboratory blood tests to determine prothrombin fragments F1+2 in blood of COPD patients

SUMMARY:
To access the clinical usefulness of F1+2 in the diagnosis of PE in patients with AECOPD who require hospitalization. Specifically, to determine whether F1+2 may have an additional value in the subgroup of patients with an abnormal D-dimer,to determine whether it may increase the proportion of patients in whom PE can be safely ruled out and to determine the sensitivity, specificity and NPV of F1+2 at various cut-off values.

ELIGIBILITY:
Inclusion Criteria:

* COPD exacerbation
* Able to give informed consent
* Able to perform spirometry

Exclusion Criteria:

* Known malignancy
* Known hypercoagulable state
* Receiving anticoagulant treatment
* Pregnancy
* Renal failure
* Allergy to iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital due to COPD exacerbation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value of Prothrombin Fragment F1+2 | Six months
  Blood test to determine predictive value of Prothrombin Fragment F1+2 in PE diagnosis in hospitalized COPD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel